CLINICAL TRIAL: NCT05309616
Title: Effects of IL-17A Inhibition on Idiopathic Subglottic Stenosis
Brief Title: Effects of Interleukin (IL)-17A Inhibition on Idiopathic Subglottic Stenosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Lilly PharmaceuticalCompany (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000031202; No NIH funding (Other: 11.09.23)
Record Dates: First submitted 2022-02-24; First posted 2022-04-04 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Idiopathic Subglottic Stenosis
Keywords: IL-17a inhibition
MeSH Terms: conditions — Idiopathic subglottic tracheal stenosis | interventions — ixekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Talz (Experimental): All participants receive Talz
  Interventions: Drug: Taltz

INTERVENTIONS:
Drug: Taltz — Participants will receive160 mg (two 80 mg injections) at week 0, followed by 80 mg at weeks 2,4,6,8,10,12 and then 80 mg every 4 weeks
  Other Names: Ixekizumab

SUMMARY:
The purpose of this phase 2 study is to examine if inhibiting IL-17A activation using the biologic drug Taltz, in idiopathic subglottic stenosis patients will decrease scar fibroblast proliferation therefore reducing or eliminating the need for invasive or repeat surgeries.

DETAILED DESCRIPTION:
The purpose of this phase 2 study is to examine if inhibiting IL-17A activation using the biologic drug Taltz, in idiopathic subglottic stenosis patients will decrease scar fibroblast proliferation therefore reducing or eliminating the need for invasive or repeat surgeries. Inhibition of the IL-17A pathway can slow or reverse the inflammation causing airway narrowing in patients with idiopathic subglottic stenosis. This would have a significant impact on quality of life for patients living with this diagnosis as it may help them to avoid frequent surgical procedures, recoveries and associated costs.

This is a single arm, open-label study where all participants will receive drug. The study population is patients with a documented diagnosis of idiopathic subglottic stenosis who are followed at Yale New Haven Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* diagnosis of idiopathic subglottic stenosis

Exclusion Criteria:

* History of active or latent tuberculosis infection
* History of inflammatory bowel disease
* Pregnancy or lactation
* Known allergic reactions to study drug
* Disease involving the vocal cords
* Individuals who are taking drugs known to trigger angioedema, including use acquired angioedema from drugs such as ACE inhibitors (e.g. Lisinopril) and nonsteroidal anti-inflammatory drugs (NSAIDs) and individuals with a history of other forms of angioedema such as hereditary and Clesterase deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of weeks between operative interventions | From baseline up to 12 months.
  The number of weeks between operative interventions will be counted. Intervention is performed once stenosis related symptoms interfere with daily life. Participants intervals will be compared to their own baseline and national databases (pre-treatment) to assess if IL-17A inhibition prolongs the interval between interventions with prolonged intervals indicating a slower progression to re-stenosis.

SECONDARY OUTCOMES:
Change in degree of stenosis measured by in-office laryngoscopy | Every 12 weeks up to 12 months
  Change in degree of stenosis measured by in-office laryngoscopy will be assessed qualitatively every 6 weeks. Degree of stenosis will be assessed as Mild, Moderate or Severe.
Change in European Quality of Life-Five Dimensions (EQ-5D) Questionnaire | Every 12 weeks up to 12 months
  EQ-5D is a standardized measure of health-related quality of life simple, generic questionnaire. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Change in RAND 36-Item short form health-related quality of life survey | Every 12 weeks up to 12 months
  The RAND-36 (SF-36) is the most widely used measure of health-related quality of life survey. It is comprised of 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions.
  Scoring the RAND 36-Item Health Survey is a two-step process. First, all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. Second, items in the same scale are averaged together to create the 8 scale scores.
Change in Clinical Chronic Obstructive Pulmonary Disease (COPD) Questionnaire (CCQ) | Every 12 weeks up to 12 months
  The CCQ consists of three subdomains: symptoms, functional state and mental state. Items are scored on a Likert scale (range 0-60). The final score is the sum of all items divided by 10; separate scores for all three domains can be calculated. Higher scores indicate a worse health status
Change in Airway, Dyspnea, Voice, and Swallowing (ADVS) Summary Assessment | Every 12 weeks up to 12 months
  A disease-specific Patient-Reported Outcome Measure validated surveys Consists of four domains (airway, dyspnea, voice and swallowing) each scored on 4 point Likert scales of functioning. This summary scale will be used to measure efficacy.
Change in Pulmonary function tests (PFT): peak expiratory flow rate in liters/second | Weekly up to 12 months
  Peak expiratory flow rate measures the maximum speed of expiration using a hand held monitor. Patients perform at home PFT weekly and report scores to the study team. Values that are 80 to 100 percent of the normal predicted peak flow readings indicate good lung function.
Change in PFT: forced expiratory flow rate in liters/second | Weekly up to 12 months
  Forced expiratory flow rate measures the volume of air that can forcibly be blown out in first 1 second, after full inspiration, using a hand held monitor. Patients perform at home PFT weekly and report scores to the study team. Values that are 80 to 120 percent of the normal predicted peak flow readings indicate good lung function.
Change in PFT: peak inspiratory flow rate in liters/second | Weekly up to 12 months
  Peak inspiratory flow rate measures the maximal flow rate obtained during an inspiratory maneuver using a hand held monitor. Patients perform at home PFT weekly and report scores to the study team. Values that are >60 L/min indicate good lung function.

CONTACTS AND LOCATIONS:
Overall Officials: Nwanmegha Young, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No